CLINICAL TRIAL: NCT05834712
Title: A Randomized, Controlled, Phase II Clinical Study on the Improvement of Malnutrition in Patients With Stage III-IVa Nasopharyngeal Carcinoma With or Without the Use of Mobile Medical Platform Full-course Nutritional Intervention
Brief Title: Patients With Stage III-IVa Nasopharyngeal Carcinoma With or Without a Mobile Medical Platform Full-course Nutritional Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-FXY-332
Record Dates: First submitted 2022-04-18; First posted 2023-04-28 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2023-08

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; mobile platform; nutritional intervention; radiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mobile Platform Intervention Group (Experimental): The mobile platform is used to evaluate the nutrition of patients 2 weeks after the first course of induction chemotherapy, before radiotherapy, during radiotherapy, after radiotherapy, and 1 month after radiotherapy. The doctor pushes individualized nutrition education, oral advice, medication advice, etc. .
  Interventions: Device: mobile platform or not mobile platform
- Non-mobile Platform Intervention Group (Active Comparator): Nutritional assessment of patients was performed at 2 weeks after 1 course of induction chemotherapy, before radiotherapy, during radiotherapy, at the end of radiotherapy, and at 1 month after the end of radiotherapy.
  Interventions: Device: mobile platform or not mobile platform

INTERVENTIONS:
Device: mobile platform or not mobile platform — Intervention using WeChat

SUMMARY:
To study the difference in the proportion of patients with nasopharyngeal carcinoma who lost more than 10% of their body weight within 1 month after radiotherapy and chemotherapy using the mobile platform for whole-process individualized nutritional rehabilitation management compared with conventional nutritional rehabilitation management.

ELIGIBILITY:
Inclusion Criteria:

* 1.Voluntarily participate and sign the informed consent in writing.
* 2.Stage III-IVa (AJCC 8th edition staging) .
* 3.Received induction chemotherapy + concurrent chemoradiotherapy .
* 4.18-70 years old.
* 5.Pathologically diagnosed with non-keratinizing nasopharyngeal carcinoma (differentiated or undifferentiated, that is, WHO type II or III).
* 6.No previous anti-tumor therapy .
* 7.ECOG score 0-1.
* 8.Ensure contraception during the study period.
* 9.Hemoglobin (HGB) ≥90 g/L, white blood cell (WBC) ≥4×109/L, platelet (PLT) ≥100×109/L.
* 10. Liver function: ALT, AST < 2.5 times the upper limit of normal (ULN), total bilirubin < 2.0 × ULN.
* 11. Renal function: serum creatinine <1.5×ULN.
* 12.Able and willing to use a mobile phone or tablet to fill in the electronic scale.

Exclusion Criteria:

* 1.Received antitumor therapy in the past.
* 2. The pathology was keratinizing squamous cell carcinoma (WHO type I).
* 3.Pregnant women who are in the reproductive period and have not taken effective contraceptive measures.
* 4. Has suffered from other malignant tumors (except for cured basal cell carcinoma or carcinoma in situ of the cervix).
* 5.Patients with significantly low heart, liver, lung, kidney and bone marrow functions.
* 6.Serious, uncontrolled medical diseases and infections.
* 7.Concurrent use of other experimental drugs or other clinical trials.
* 8. Refused or unable to sign the informed consent to participate in the trial.
* 9.Those who have other contraindications to treatment.
* 10.Persons with personality or mental disorders, no capacity for civil conduct or limited capacity for civil conduct.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2023-09-24 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
weight loss | 1 month after chemoradiotherapy
  Differences in the proportion of patients who lost >10% of their body weight at 1 month after chemoradiotherapy between experimental and control groups

SECONDARY OUTCOMES:
weight loss >10% | at the end of chemoradiotherapy
  Differences in the proportion of patients who lost >10% of their body weight at the end of chemoradiotherapy between experimental and control groups
weight loss >20% | at the end of chemoradiotherapy
  Differences in the proportion of patients who lost >20% of their body weight at the end of chemoradiotherapy between experimental and control groups
ncidence rate of adverse events (AEs) | at the end of chemoradiotherapy
  Analysis of acute and late adverse events (AEs) are evaluated. Numbers of patients of treatment-related adverse events(acute toxicity) as assessed by CTCAE v5.0.Numbers of patients of late radiation toxicities were assessed using the Radiation Therapy Oncology Group and European Organization for Research and Treatment of Cancer late radiation morbidity scoring scheme.
change of PG-SGA | 1 month after chemoradiotherapy
  Scored Patient-Generated Subjective Global Assessment (PG-SGA).It consists of two parts: the patient's self-assessment part and the medical staff's assessment part. The specific contents include seven aspects, including body weight, food intake, symptoms, activity and physical function, the relationship between disease and nutritional needs, metabolic needs, and physical examination. The first 4 Each aspect is evaluated by the patient himself, and the last three aspects are evaluated by the medical staff. The overall evaluation includes qualitative evaluation and quantitative evaluation.
change of NRS2002 | 1 month after chemoradiotherapy
  The outstanding advantage of NRS2002 is that it can predict the risk of malnutrition, and can proactively and dynamically judge the changes in the nutritional status of patients, which is convenient for timely feedback of the nutritional status of patients, and provides evidence for adjusting nutritional support programs. It is a better nutritional risk screening tool.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nasopharyngeal Carcinoma, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No